CLINICAL TRIAL: NCT06347094
Title: Precision Nutrition to Improve Cardiometabolic Health With Dietary (Poly)Phenols (PRE-CARE-DIET)
Brief Title: Precision Nutrition to Improve Cardiometabolic Health With Dietary (Poly)Phenols
Acronym: PRE-CARE-DIET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other); University of Milan (Other); Foundation for Liver Research (Other); National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Pedro M. Mena Parreño, PhD, University of Parma
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 610/2023/SPER/UNIPR
Record Dates: First submitted 2024-03-04; First posted 2024-04-04 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Individual Variability in (Poly)Phenol Metabolism; Cardiometabolic Health; Personalized Dietary Intervention; Obesity
Keywords: nutritional intervention study; personalized nutrition; cardiometabolic risk; obesity; (poly)phenols; metabotypes; inter-individual variability; food-gut-host interactions; predictive models
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Metabotypes will also be masked to participants and investigators, while the dietary treatment will not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metabotype X, Treatment (Experimental): Subjects belonging to a specific aggregate phenolic metabotype (X) to which a diet with an increase of 50% in the actual (poly)phenol intake will be given, through personalized dietary plans.
  Interventions: Other: Personalized Dietary Plan; Dietary Supplement: Oral (Poly)phenol Challenge Test (OPCT)
- Metabotype X, Control (Experimental): Subjects belonging to a specific aggregate phenolic metabotype (X) to which general dietary recommendations for a healthy diet will be given.
  Interventions: Dietary Supplement: Oral (Poly)phenol Challenge Test (OPCT); Other: General Dietary Advice
- Metabotype Y, Treatment (Experimental): Subjects belonging to a specific aggregate phenolic metabotype (Y) to which a diet with an increase of 50% in the actual (poly)phenol intake will be given, through personalized dietary plans.
  Interventions: Other: Personalized Dietary Plan; Dietary Supplement: Oral (Poly)phenol Challenge Test (OPCT)
- Metabotype Y, Control (Experimental): Subjects belonging to a specific aggregate phenolic metabotype (X) to which general dietary recommendations for a healthy diet will be given.
  Interventions: Dietary Supplement: Oral (Poly)phenol Challenge Test (OPCT); Other: General Dietary Advice

INTERVENTIONS:
Other: Personalized Dietary Plan — Prescription of dietary plans increasing the intake of (poly)phenols through consumption of foods rich in these compounds, in the context of a balanced, personalised diet
  Arms: Metabotype X, Treatment; Metabotype Y, Treatment
Dietary Supplement: Oral (Poly)phenol Challenge Test (OPCT) — Nutritional challenge with standardized (poly)phenol-rich tablets
Other: General Dietary Advice — Prescription of balanced dietary plans
  Arms: Metabotype X, Control; Metabotype Y, Control

SUMMARY:
This chronic study aims at assessing whether the effects of a personalized, plant-based diet rich in (poly)phenols on cardiometabolic health depend on the capability to metabolize dietary (poly)phenols, creating predictive models able to explain, at individual level, the cardiometabolic response. This study presents an observational part, for targeted recruitment and volunteers characterization, and an experimental part for the dietary and deep phenotyping.

DETAILED DESCRIPTION:
The recruitment will be carried out to prospectively include 330 subjects belonging to two aggregate phenolic metabotypes, that will be compared in the intervention part (1:1). To do so, a maximum of 500 subjects at cardiometabolic risk will be screened following an oral (poly)phenol challenge test (OPCT). In the observational phase, eating habits and lifestyle data will be collected, and these will serve as a run-in for the experimental phase. In the experimental phase, two-thirds of the participants within each metabotype will be randomly allocated to the treatment arm: 50% increase in the (poly)phenol intake, with a minimum daily intake of 500 mg. Treatment allocation shifts minimally the dietary habits of treated participants to allow causal explanations. No changes in the (poly)phenol intake will be asked to the control arm, composed of one-third of the subjects in each metabotype. Blood pressure and heart rate will also be measured and anthropometric data collected. Information will be accessed on cardiometabolic risk scores, cardiometabolic health biomarkers, inflammatory markers, hormones, metabolism of food components, genetic polymorphisms, gut and saliva microbiota profile, etc., through the collection of saliva, urine, blood, and stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Adults (40-80 y.o.)
* Non-clinically diagnosed for cardiometabolic diseases at baseline examination
* At least one of the following risk factors: overweight or obese, central obesity (waist:hip ratio > 0.90 in males and > 0.85 in females or waist circumference ≥ 94 cm in males and ≥ 80 cm in females), hypertension (systolic BP > 130 or diastolic BP > 85 mm Hg), low high-density lipoprotein cholesterol levels (< 40 mg/dL (1.03 mmol/L) in males, < 50 mg/dL (1.29 mmol/L) in females), or elevated total cholesterol (≥ 200 mg/dL), low-density lipoprotein cholesterol (≥ 130 mg/dL (4.1 mmol/L)), triglyceride (> 150 mg/dL (1.7 mmol/L)), fasting glucose (> 100 mg/dL (5.6 mmol/L)) levels, or microalbuminuria (urinary albumin excretion ratio ≥ 20 μg/min or albumin:creatinine ratio ≥ 30 mg/g).

Exclusion Criteria:

* BMI < 18.5 or > 34.9 kg/m²
* Past cardiovascular events and metabolic diseases including diabetes
* Inflammatory bowel diseases or gastro-intestinal surgery (other than appendectomy)
* Cholecystectomy within the past 5 years
* Renal or hepatic diseases
* Levels of estimated Glomerular Filtration (eGFR) < 60 mL/min/1.73 m²
* Aspartate transaminase (AST)/alanine aminotransferase (ALT) 2.5 times the upper limits of normal
* Immunodeficiency or autoimmune diseases (other than well-compensated hypothyroidism)
* Mental disorders
* Hormone therapy (other than that used for hypothyroidism, birth-control or menopause symptoms)
* Antibiotic therapy within the last month before the study
* Food allergies associated with the consumption of plant foods or foods that will be provided in the study
* Difficulties or major inconveniences in changing dietary habits or adhering to a plant-based Mediterranean-type diet
* Presence of chewing or swallowing disorders
* Pregnancy or lactation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing the effect of a (poly)phenol-rich diet on 10-year cardiovascular risk: Systematic Coronary Risk Estimation | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Assessing the effect of a (poly)phenol-rich diet on 10-year risk of cardiovascular disease using the Systematic Coronary Risk Estimation (SCORE2) for volunteers aged between 40 and 69 years, considering different aggregate phenolic metabotypes. Interpretation of the result depends on the patient's age as the cut-off risk levels are numerically different for various age groups: low-moderate Cardiovascular Disease (CVD) risk (< 2.5% for < 50 years; < 5% for 50-69 years), high CVD risk (2.5% to < 7.5% for < 50 years; 5% to < 10% for 50-69 years), very high CVD risk (≥ 7.5% for < 50 years; ≥ 10% for 50-69 years).
Assessing the effect of a (poly)phenol-rich diet on 10-year cardiovascular risk: Systematic Coronary Risk Estimation-Older Persons | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Assessing the effect of a (poly)phenol-rich diet on 10-year risk of cardiovascular disease using the Systematic Coronary Risk Estimation-Older Persons (SCORE2-OP) for volunteers aged between 70 and 89 years, considering different aggregate phenolic metabotypes. Interpretation of the result depends on the patient's age as the cut-off risk levels are numerically different for various age groups: low-moderate CVD risk (< 7.5% for ≥ 70 years), high CVD risk (7.5% to < 15% for ≥ 70 years ), very high CVD risk (≥ 15% for ≥ 70 years).

SECONDARY OUTCOMES:
Anthropometric measurements: weight, height and body mass index | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Weight (measured in kilograms) and height (measured in meters) will be assessed using a balance and a stadiometer, respectively. These measures will be combined to report the Body Mass Index (BMI) using the following formula: kg/m^2.
Anthropometric measurements: waist and hip circumferences detection | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Waist circumference (measured in centimeters) and hip circumference (measured in centimeters) will be assessed using an inelastic meter. These measures will be combined to report waist-to-height ratio and waist-to-hip ratio using the following formulas: waist circumference (cm)/height (cm) and waist circumference (cm)/hip circumference (cm), respectively.
Body composition: bioelectrical impedance analysis | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Body composition estimation will be assessed using a bioelectrical impedance analysis (BIA). It is a tool that provides an estimate of qualitative and quantitative analysis of body composition and distribution.
Blood pressure | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Systolic and diastolic blood pressure measured in millimeters of mercury (mmHg) of each volunteer will be obtained after a 5-min rest in a seated position.
Heart rate | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Heart rate, measured in beats per minute (bpm) of each volunteer will be obtained after a 5-min rest in a seated position.
Biomarkers of cardiometabolic health: hematochemical and urine analysis | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Blood samples will be collected for the assessment, measured in milligrams per deciliter, of total cholesterol (mg/dL), HDL-cholesterol (mg/dL), triglycerides (mg/dL), glucose (mg/dL), lipoprotein a (mg/dL), apolipoprotein A1 (mg/dL), apolipoprotein B (mg/dL) and uric acid (mg/dL).
Biomarkers of cardiometabolic health: alanine aminotransferase, aspartate aminotransferase and gamma glutamyl transferase | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Blood samples will be collected for the assessment, measured in enzymatic unit activity per liter, of alanine aminotransferase (U/L), aspartate aminotransferase (U/L) and gamma glutamyl transferase (U/L).
Biomarkers of cardiometabolic health: homocysteine | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Homocysteine, measured in milligrams per liter, will be assessed from serum samples.
Biomarkers of cardiometabolic health: insulin | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Insulin, measured in micro Insulin Units per milliliter, will be assessed from plasma samples.
Biomarkers of cardiometabolic health: glycated hemoglobin and glycated albumin | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Blood samples will be collected for the assessment, measured in percentage of total hemoglobin, of glycated hemoglobin (HbA1c (%)) and glycated albumin (%).
Biomarkers of cardiometabolic health: quantitative insulin-sensitivity check index | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Fasting insulin sensitivity will be estimated through the quantitative insulin-sensitivity check index (QUICKI) using the following formula: 1/log(fasting insulin (uUI/mL)) + log(fasting glucose (mg/dL)).
Biomarkers of cardiometabolic health: homeostasis model assessment beta-cell function | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Insulin secretion capacity will be estimated through the homeostasis model assessment beta-cell function (HOMA-β) index using the following formula: 360 * insulin (uUI/mL)/glucose (mg/dL) - 55.
Biomarkers of cardiometabolic health: homeostasis model assessment of insulin resistance | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Insulin resistance will be estimated through the homeostasis model assessment of insulin resistance (HOMA-IR) index using the following formula: glucose (mg/dL) * insulin (uUI/mL)/82 * 7.
Inflammatory status | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Plasma samples will serve to determinate the inflammatory status monitoring specific cytokines (Tumor Necrosis Factor α, InterLeukin-1β, InterLeukin-6, InterLeukin-8, InterLeukin-10, and Monocyte Chemoattractant Protein-1), adhesion molecules (Vascular cell adhesion protein-1, Intercellular Adhesion Molecule-1, E-selectin), and high sensitivity C reactive protein (hsCRP), using a customized magnetic bead-based multiplex assays.
Risk prediction scores: Framingham General Cardiovascular Risk Score - 10-years | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Framingham General Cardiovascular Risk Score (FRS) - 10 years will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. The FRS estimates the 10-years risk of manifesting clinical CVD (CAD, Stroke, cardiac death). Risk is considered low if the FRS is less than 10%, moderate if it is 10% to 19%, and high if it is 20% or higher.
Risk prediction scores: Framingham General Cardiovascular Risk Score - 30-years | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Framingham General Cardiovascular Risk Score (FRS) - 10 years will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. The FRS estimates the 30-years risk of manifesting clinical CVD (CAD, Stroke, cardiac death). Risk is considered low if the FRS is less than 12%, moderate if it is 12% to 40%, and high if it is 40% or higher.
Risk prediction scores: Hard Coronary Heart Disease - 10-years risk | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Framingham Heart Study Primary Risk Functions for Hard Coronary Heart Disease (HCHD) 10-year risk will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. The HCHD estimates the 10-years risk of manifesting myocardial infarction or coronary death. Risk is considered low if the HCHD is less than 1%, moderate if it is 1%, and high if it is 2% to 11% for female; risk is considered low if the HCHD is less than 1%, moderate if it is 1%, and high if it is 2% to 25% for male.
Risk prediction scores: First Coronary Heart Disease - 2-years risk | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Framingham Heart Study Primary Risk Functions for First Coronary Heart Disease (2-years risk) will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. This risk score estimates the 2-years risk of manifesting a first event of myocardial infarction or coronary death. Risk is considered low if the score is less than 0%, moderate if it is 0% to 1%, and high if it is 1% or higher for female; risk is considered low if the score is less than 0%, moderate if it is 0% to 1%, and high if it is 1% to 6% for male.
Risk prediction scores: Framingham Heart Study for Diabetes | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Framingham Heart Study Primary Risk Functions for Diabetes will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. This risk score estimates the risk of manifesting type 2 diabetes mellitus (fasting blood glucose at or above 126 mg/dL) in 8 years. Risk is considered low if the score is less than 3% and high if it is 4% to 18%.
Risk prediction scores: Framingham Heart Study for Hypertension | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Framingham Heart Study Primary Risk Functions for Hypertension will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. This risk score estimates the risk of incidence of hypertension. Risk is considered low if the score is less than 5%, moderate if it is 5% to 10%, and high if it is higher than 10%.
Risk prediction scores: Framingham Heart Study for Stroke | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Framingham Heart Study Primary Risk Functions for Stroke will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. This risk score estimates the 10-year probability of stroke. The risk score is given as a percentage and higher percentage values correspond to an increased risk of stroke.
Risk prediction scores: Framingham Heart Study for Fatty Liver Disease | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Framingham Heart Study Primary Risk Functions for Fatty Liver Disease will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. This risk score estimates the 10-year risk of CVD events in individuals with non-alcoholic fatty liver disease (NAFLD) The risk score is given as a percentage and higher percentage values correspond to an increased risk of CVD events.
Risk prediction scores: Atherosclerotic Cardiovascular Disease | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Atherosclerotic Cardiovascular Disease (ASCVD) risk will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. It is an index of the 10-year risk of having a cardiovascular problem, such as a heart attack or stroke. The ASCVD risk score is given as a percentage and there are four groupings: a 0 to 4.9 percent risk is considered low; a 5 to 7.4 percent risk is considered borderline; a 7.5 to 20 percent risk is considered intermediate; a greater than 20 percent risk is considered high.
Risk prediction scores: QRESEARCH risk estimator version 3 | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The QRESEARCH risk estimator version 3 (QRISK3®) will be assessed to understand their relationship with the aggregate phenolic metabotypes observed. It is an index of the 10-year risk of having a cardiovascular problem, such as a heart attack or stroke. The QRISK3® risk score is given as a percentage and there are three groupings: low risk if the QRISK3 score of less than 10%; moderate risk if the QRISK3 of 10-20%; high risk if the QRISK3 score of more than 20%.
Risk prediction scores: QDiabetes Score | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The QDiabetes Score® will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. QDiabetes® is a validated tool which predicts the absolute risk of developing type 2 diabetes in the next 10 years. The QDiabetes Score® risk score is given as a percentage: high risk is defined for QDiabetes of 5.6% or greater, while it is low for lower values.
Risk prediction scores: Finnish Diabetes Risk Score | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Finnish Diabetes Risk Score (FINDRISC) will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. FINDRISC is a prediction tool to identify patients at risk of developing diabetes. A risk score of 0-14 points indicates a low to moderate risk of diabetes (1-17% chance of diabetes over 10 years). A risk score of 15-20 points indicates a high risk of diabetes (33% chance of diabetes over 10 years). A risk score of >20 points indicates a very high risk of diabetes (50% chance of diabetes over 10 years).
Risk prediction scores: Cuore Project - Calculating the individual risk score | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  The Calculating the individual risk score (Italian CVD risk score) will be assessed to understand the relationship with the aggregate phenolic metabotypes observed. Six cardiovascular risk categories were constructed, called MCV (from I to VI): the MCV risk category indicates how many persons out of 100 with the same characteristics will fall ill over next 10 years. Risk is considered: below 5% for MCV I; 5% to 10% for MCV II; 10% to 15% for MCV II; 15% to 20% for MCV IV; 20% to 30% for MCV V; over 30% for MCV VI
Evaluation of adherence to healthy and sustainable dietary models: the Healthy Eating Index | Visit 2 (after 4 weeks from the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Adherence to healthy dietary patterns will be assessed by the Healthy Eating Index (HEI), which is a measure of diet quality used to assess how well a set of foods aligns with key recommendations and dietary patterns. The HEI uses a scoring system from 0 to 100. There are two groupings: 1) "Adequacy components" represent the food groups, subgroups, and dietary elements that are encouraged and for these components, higher scores reflect higher intakes, because higher intakes are desirable; 2) "Moderation components" represent the food groups and dietary elements for which there are recommended limits to consumption and for moderation components, higher scores reflect lower intakes, because lower intakes are more desirable.
Evaluation of adherence to healthy and sustainable dietary models: Italian Mediterranean Index | Visit 2 (after 4 weeks from the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Adherence to Italian Mediterranean diet will be assessed by the Italian Mediterranean Index. The score is calculated from intake of 11 items: high intakes of six typical Mediterranean foods (pasta, typical Mediterranean vegetables, fruit, legumes, olive oil and fish; low intakes of four "non-Mediterranean" foods (soft drinks, butter, red meat and potatoes); and alcohol. If consumption of typical Mediterranean foods is in the 3rd tertile of the distribution, the person receives 1 point; all other intakes receive 0 points. If consumption of non-Mediterranean foods is in the first tertile of the distribution the person receives 1 point. Alcohol receives 1 point for intake up to 12 g/day; abstainers and persons who consume >12 g/day receive 0. Possible scores range from 0 to 11.
Evaluation of adherence to healthy and sustainable dietary models: Greek Mediterranean Index | Visit 2 (after 4 weeks from the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  To evaluate the adherence to and healthy and sustainable dietary, the Greek Mediterranean Index will be assessed with a nine-point score for the consumption of vegetables, legumes, fruit and nuts, cereal, ﬁsh, meat,dairy, alcohol, and lipids. Using the sex-speciﬁc median, a value of 0 will be given to participants whose consumption of vegetables, legumes, fruits and nuts, cereals, and ﬁsh is below the median consumption, while a value of 1 will be assigned in the opposite case. Study participants with a below-median consumption of meat and dairy products will be assigned a value of 1, whereas a value of 0 will be given to those with an above-median consumption. For ethanol, men consuming 10-50 g/day and women consuming 5-25 g/day will be given a value of 1. The score is categorized into three categories: low adherence, including individuals with a total score of 0 to 3 points; intermediate adherence, with a score of 4 to 5 points; and high adherence,with a score of 6 to 9 points.
Evaluation of adherence to healthy and sustainable dietary models: DASH Index | Visit 2 (after 4 weeks from the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Adherence to healthy dietary patterns will be assessed by the Dietary Approaches to Stop Hypertension (DASH) Index.
  The DASH Index is comprised of 8 components (7 food groups and one nutrient). The scoring system is based on quintile rankings; for intakes of fruit (includes fruit juice), vegetables (excludes potatoes), low-fat dairy products, whole grains, and nuts, seeds, and legumes, individuals receive a score from 1 (lowest quintile) to 5 (highest quintile). In contrast, individuals receive a score from 1 (highest quintile) to 5 (lowest quintile) for intakes of sodium, sugar-sweetened beverages, and red and processed meat. Men and women are classified into quintiles separately. Component scores are summed to a total DASH score that ranges from a minimum of 8 to a maximum of 40 points.
Evaluation of adherence to Mediterranean diet | Visit 2 (after 4 weeks from the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Adherence to Mediterranean Diet will be assessed through the MEDI-Lite questionnaire.
Nutritional and energy assessment: LARN | Visit 2 (after 4 weeks from the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Nutritional and energy requirements will be assessed considering the "Reference Intake Levels of Nutrients and Energy for the Italian Population for the Italian population" (LARN) recommendation using dietary records.
Nutritional and energy assessment: EPIC | Visit 2 (after 4 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Nutritional and energy requirements will be assessed through the food frequency questionnaire European Prospective Investigation into Cancer and Nutrition (EPIC).
Dietary intake assessment of plant bioactive compounds and dietary components related to gut microbiome | Visit 2 (after 4 weeks from the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  (Poly)phenol intake will be estimated using a food database. The same methodology will serve to calculate the intake of other plant bioactive compounds and dietary components associated with the gut microbiome, by matching food frequency questionnaires, and the dietary records data with databases.
Lifestyle factors assessment: general information | Visit 1 (beginning of the study), Visit 2 (4 weeks after the beginning of the study) Visit 3 (8 weeks after the beginning of the study), Visit 4 (16 weeks after the beginning of the study) and Visit 5 (24 weeks after the beginning of the study)
  General information, such as age, sex, smoking habits, childbirth, breastfeeding, will be assessed through an enrollment questionnaire.
Lifestyle factors assessment: sleep quality (PSQI) | Visit 1 (beginning of the study), Visit 2 (4 weeks after the beginning of the study) Visit 3 (8 weeks after the beginning of the study), Visit 4 (16 weeks after the beginning of the study) and Visit 5 (24 weeks after the beginning of the study)
  Assessing the contribution of sleep quality through the questionnaire Pittsburgh Sleep Quality Index (PSQI). Scoring of answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme. A global sum of "5" or greater indicates a "poor" sleeper, while an overall sum of less than "5" indicates a "good" sleeper.
Lifestyle factors assessment: sleep quality (ESS) | Visit 1 (beginning of the study), Visit 2 (4 weeks after the beginning of the study) Visit 3 (8 weeks after the beginning of the study), Visit 4 (16 weeks after the beginning of the study) and Visit 5 (24 weeks after the beginning of the study)
  Assessing the contribution of sleep quality through the questionnaire Epworth Sleepiness Scale (ESS). The test is a list of eight situations in which it is rate the tendency to become sleepy on a scale of 0 to 3: 0 (no chance of dozing), 1 (slight chance of dozing), 2 (moderate chance of dozing), and 3 (high chance of dozing). The total ESS score is based on a scale of 0 to 24 and can be interpreted as follows: 0-5 Lower Normal Daytime Sleepiness; 6-10 Higher Normal Daytime Sleepiness; 11-12 Mild Excessive Daytime Sleepiness; 13-15 Moderate Excessive Daytime Sleepiness; 16-24 Severe Excessive Daytime Sleepiness
Lifestyle factors assessment: sleep quality (ISI) | Visit 1 (beginning of the study), Visit 2 (4 weeks after the beginning of the study) Visit 3 (8 weeks after the beginning of the study), Visit 4 (16 weeks after the beginning of the study) and Visit 5 (24 weeks after the beginning of the study)
  Assessing the contribution of sleep quality through the questionnaire Insomnia Severity Index (ISI).
Lifestyle factors assessment: physical activity (IPAQ) | Visit 1 (beginning of the study), Visit 2 (4 weeks after the beginning of the study) Visit 3 (8 weeks after the beginning of the study), Visit 4 (16 weeks after the beginning of the study) and Visit 5 (24 weeks after the beginning of the study)
  Assessing the contribution of physical activity through the questionnaire International Physical Activity Questionnaire (IPAQ).
Lifestyle factors assessment: state of health (BDI) | Visit 1 (beginning of the study), Visit 2 (4 weeks after the beginning of the study) Visit 3 (8 weeks after the beginning of the study), Visit 4 (16 weeks after the beginning of the study) and Visit 5 (24 weeks after the beginning of the study)
  Assessing the contribution of state of health through the questionnaire Beck's Depression Inventory (BDI).
Lifestyle factors assessment: state of health (SF-36) | Visit 1 (beginning of the study), Visit 2 (4 weeks after the beginning of the study) Visit 3 (8 weeks after the beginning of the study), Visit 4 (16 weeks after the beginning of the study) and Visit 5 (24 weeks after the beginning of the study)
  Assessing the contribution of state of health through the questionnaire Short Form Health Survey 36 (SF-36).
(Poly)phenol metabolites and changes in the prevalence of aggregate phenolic metabotypes | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  True internal exposure to dietary (poly)phenols will be assessed by analysing the circulating metabolites of (poly)phenols in the plasma, urine, and faecal samples collected. Validated targeted ultra performance liquid chromatography method coupled with triple quadrupole mass spectrometry (UPLC-QqQ-MS/MS) and untargeted Ultra Performance Liquid Chromatography-Ion Mobility Spectrometry-High-Resolution Mass Spectrometry (UPLC-IMS-HRMS) methods will be used.
Other plant bioactive metabolites | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  True internal exposure to plant bioactive compounds will be assessed by analysing the circulating plant bioactive compounds (carotenoids, phytosterols, alkaloids (mainly purines and pyridines), thiosulfinates, and alkylresorcinols), in the plasma, urine, and faecal samples collected. Validated targeted ultra performance liquid chromatography method coupled with triple quadrupole mass spectrometry (UPLC-QqQ-MS/MS) and untargeted Ultra Performance Liquid Chromatography-Ion Mobility Spectrometry-High-Resolution Mass Spectrometry (UPLC-IMS-HRMS) methods will be used.
Food/gut/host-derived metabolites | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Metabolites playing a role in the diet-gut microbiome-host interactions will be evaluated in plasma/urine/faeces samples using targeted ultra performance liquid chromatography method coupled with triple quadrupole mass spectrometry (UPLC-QqQ-MS/MS) and untargeted Ultra Performance Liquid Chromatography-Ion Mobility Spectrometry-High-Resolution Mass Spectrometry (UPLC-IMS-HRMS) methods. Main compounds to be targeted are short-chain fatty acids, L-carnitine, choline, phosphatidylcholine, trimethylamine, trimethylamine N-oxide, tryptophan and indole derivatives, phenylalanine and phenylacetate, tyrosine derivatives, 4-ethylphenylsulfate, p-cresol-sulfate, and primary and secondary bile acids.
Biomarkers of food intake and of healthy dietary patterns | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Multiple metabolites associated with the consumption of food groups and foodstuffs will be analysed in urine samples and, in case, in plasma, using ultra performance liquid chromatography method coupled with triple quadrupole mass spectrometry (UPLC-QqQ-MS/MS) methods, to provide objective information on participants' diet. Moreover, a comprehensive panel of biomarkers related to healthy dietary patterns will be analysed in plasma/urine samples by using Ultra-performance liquid chromatography-mass spectrometry (UPLC-MS) methods procedures reported in literature.
Untargeted metabolomics | Visit 1 (at the beginning of the study), Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Urine/plasma/fecal samples will be subjected to untargeted Liquid Chromatography-Ion Mobility Spectrometry-Mass Spectrometry (LC-IMS-MS) metabolomics approach to assess potential differences among the metabolomes of individuals belonging to different aggregate phenolic metabotypes.
Genetic differences | Visit 3 (after 8 weeks from the beginning of the study)
  Genotyping will be conducted using genome wide, single nucleotide polymorphisms (SNPs) array approach untargeted methodology, using commercially available SNPs. Genomic DNA will be prepared from blood samples.
Gut microbiota composition | Visit 3 (after 8 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  Microbial profiling in faeces samples will be carried out by an internal transcribed spacer (ITS)-based method for cataloguing of bacterial communities at (sub)species level.
Oral microbiota composition | Visit 5 (after 24 weeks from the beginning of the study)
  Microbial profiling in saliva samples will be carried out by an internal transcribed spacer (ITS)-based method for cataloguing of bacterial communities at (sub)species level.
Biomarkers of adipose tissue function | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  A panel of biomarkers related to the adipose tissue function (adiponectin, leptin, and resistin) will be evaluated in plasma samples.
Biomarkers of food intake regulation | Visit 3 (after 8 weeks from the beginning of the study), Visit 4 (after 16 weeks from the beginning of the study) and Visit 5 (after 24 weeks from the beginning of the study)
  A panel of biomarkers related to food intake regulation (ghrelin, glucagon-like peptide 1, cholecystokinin, gastric inhibitory peptide) will be analysed in plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro M Mena Parreño, PhD, Principal Investigator — University of Parma
Locations (2):
- Italy (2):
  - University of Parma - Plesso Biotecnologico Integrato, Parma, PR
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR

IPD SHARING:
Plan to Share IPD: No